CLINICAL TRIAL: NCT01495689
Title: A Pilot Randomized Control Trial of Smoking Cessation Using The Ottawa Model With the SmartCard in Out-patient Respirology Clinic Setting
Brief Title: Smoking Cessation With the Ottawa Model and SmartCard in Out-patient Respirology Clinic Setting
Acronym: Quit&Win
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Smita Pakhale, Associate Scientist and Assistant Professor, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHRI
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; respirology Out-patient setting; SmartCard
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Usual care for smoking cessation will be delivered to the control arm which comprises of strong physician advice, brief counseling from the clinic nurse +/- a prescription for smoking cessation aid if requested and willing
  Interventions: Behavioral: Usual care
- Ottawa Model with SmartCard (Experimental): On-site counseling for Smoking Cessation along with the IVR automated telephone call follow-up and SmartCard worth $110 towards purchase of smoking cessation aids
  Interventions: Behavioral: Ottawa Model with SmartCard

INTERVENTIONS:
Behavioral: Ottawa Model with SmartCard — On-site counseling for Smoking Cessation along with the IVR automated telephone call follow-up and SmartCard worth $110 towards purchase of smoking cessation aids
  Other Names: Ottawa Model of Smoking Cessation and SmartCard
  Arms: Ottawa Model with SmartCard
Behavioral: Usual care — Usual care or control arm will receive strong physician advice, brief counseling from clinic nurse +/- a prescription for smoking cessation aid if requested and willing
  Other Names: Usual care as per current practice
  Arms: Usual Care

SUMMARY:
Cigarette smoking is the most harmful and quitting smoking is very difficult. Despite quitting, it is very difficult to stay quit for long term. In Ottawa the investigators are very lucky to have designed and developed the Ottawa Model for Smoking Cessation ("Ottawa Model"). This project is an end result of pain staking research. The Ottawa Model has been implemented very successfully to the hospitalized patients and has shown very promising results of higher quitting rates.

Our objective is to modify the Ottawa Model to suit the needs of patients attending out-patient respirology clinics. The investigators aim to apply the modified Ottawa Model along with the SmartCard to the adult smokers who attend the investigators out-patient Respirology clinic at the Ottawa Hospital.

The investigators aim to train a nurse in clinical aspects and implementation of the protocols related to the Ottawa Model. The trained nurse will contact the smokers attending the clinic. Those subjects willing to participate in this study will be divided in to two groups. One group of subjects will get counseling and SmartCard on the day of the clinic and follow-up phone calls. The SmartCard is worth $110 toward the purchase of quit smoking medications (i.e. nicotine patch/gum, varenicline, or bupropion). The subjects can re-deem the card at the investigators hospital pharmacy. Those in the control group will be followed-up as the investigators are currently doing i.e. with standard smoking cessation counseling from the clinic physician and the nurse, +/- prescription for smoking cessation aids without access to the study nurse and the extra counseling or SmartCard. The investigators aim to find increased quitting rates in the group getting on-site access to the smoking cessation aids with the Smartcard and counseling.

There are no studies implementing the Ottawa Model along with the SmartCard in out-patient respirology setting so far. The Ottawa Model has proven to be very successful in the in-patient subjects. Thus, the investigators believe, the investigators can modify the Ottawa Model and make it fit the out-patient Respirology setting and increase the quitting rates.

DETAILED DESCRIPTION:
Design: Parallel group randomized control trial Method: All adult current smokers attending respirology clinic at the Ottawa General Hospital will be approached to participate. Concealed random allocation will be done if the subject is willing and signed the written informed consent. Experimental arm will receive counseling on site enrollment in the Ottawa Model of Smoking Cessation which includes IVR automated telephone follow-up and will receive a SmartCard worth $110 towards purchase of smoking cessation aids. Usual care arm will receive current usual care in our clinic i.e. strong physician advice, +/- prescription for smoking cessation aids if requested or willing.

As a priori, a third arm was added to the parent study entitled, "A PILOT IMPLEMENTATION OF BUDDHIST MINDFULNESS TRAINING COMBINED WITH THE OTTAWA MODEL FOR SMOKING CESSATION IN AN OUT-PATIENT RESPIROLOGY CLINIC SETTING". For this arm, research ethics board approval was sought and 10 participants were approached.

ELIGIBILITY:
Inclusion Criteria:

* All adult >18 years of age attending Respirology Clinic at the Ottawa General hospital
* Current smokers (anyone who had smoked any form of tobacco in the 6 months prior to the clinic visit)
* Willing to set quit dates in next 30 days

Exclusion Criteria:

* Subjects with less than 2 year life expectancy (end stage cancer, end stage lung or heart disease etc) and/or receiving palliative care
* Not willing to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smita Pakhale, MD, FRCPC, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled and randomized 49 (54.4%) of 90 respirology patients identified as smokers at their routine respirology clinic appointments between November 2011 and December 2012.
Period: Overall Study
Arm/Group | Usual Care | Ottawa Model With SmartCard
Started | 26 | 23
Completed | 16 | 16
Not Completed | 10 | 7
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Ottawa Model With SmartCard | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (10.4) | 48.3 (12.6) | 49.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 13 | 11 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Confirmed (Exhaled CO ≤ 10 Ppm) Self-reported Continuous Abstinence at 26 Weeks.
Description: The primary outcome will be measured at 26 weeks: (1) bio-chemically confirmed 7-day point prevalence abstinence; and (2) self reported continuous abstinence since randomization. Participants who will not be available for follow-up will be considered smokers. At the 26 week follow-up, all patients who report being abstinent from smoking will have their smoking status confirmed by measurement of a CO sample. If any CO will be >10 ppm, the subject will be considered a smoker.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ottawa Model With SmartCard
Number analyzed (Participants) | 26 | 23
Participants | 26 | 23

2. Primary Outcome: Self-reported Smoking Status
Description: Self-reported smoking status was the primary indicator of effectiveness and was obtained at 26-52 weeks. Participants were asked to respond "yes" or "no" to the question "Do you still smoke?"
Time Frame: 52 weeks
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ottawa Model With SmartCard
Number analyzed (Participants) | 26 | 23
Participants
  Self-reported non-smoker status | 2 | 4
  did not report report non-smoker status | 24 | 19

3. Secondary Outcome: Rate of Recruitment and Retention
Description: Rate of recruitment and retention will be evaluated which will inform feasibility of a larger trial
Time Frame: 52 weeks
Population: [not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Ottawa Model With SmartCard
Number analyzed (Participants) | 26 | 23
Participants
  Complete self-reported smoking status data | 16 | 16
  Did not complete self-reported smoking status data | 10 | 7

ADVERSE EVENTS:
Arm/Group | Usual Care | Ottawa Model With SmartCard
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

LIMITATIONS AND CAVEATS:
Small sample size is not sufficient for a statistically significant intervention effect to be detected.

Control participants were contacted monthly by the research team and were asked to set a quit date; it may be argued that this represents an enhanced version of standard care.

Financial limitations: might resulted in shorter NRT treatment than the standard of care.

Recruitment bias - we recruited low educational and income levels and the study was limited to a single site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No